CLINICAL TRIAL: NCT01153113
Title: Phase II Study of Active Immunotherapy With Mature, Human Telomerase Reverse Transcriptase Messenger RNA -Transfected, Autologous Dendritic Cells (DC) Administered In A Prime-Boost Format to Subjects With Metastatic Prostate Cancer
Brief Title: Human Telomerase Reverse Transcriptase Messenger RNA (hTERT mRNA) Transfected Dendritic Cell Vaccines
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IND has been withdrawn and the study is closed.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAMP hTERT DC Vaccine
Record Dates: First submitted 2010-03-31; First posted 2010-06-29 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-02

CONDITIONS: Metastatic Prostate Cancer
Keywords: adenocarcinoma of the prostate; metastatic prostate adenocarcinoma, Stage (T1-4, N+, M0) or (T1-4, N0-3, M+); rising PSA levels while maintained on LHRH analogues
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): • 5x106 cells per infusion administered ID
  Interventions: Biological: hTERT mRNA DC
- Treatment Arm B (Experimental): • 1x107 cells per infusion administered ID (Treatment arm B).
  Interventions: Biological: hTERT mRNA DC

INTERVENTIONS:
Biological: hTERT mRNA DC — Subjects receive 1x107 cells per infusion administered ID at study week 1, 2, 3, 4, 5, 6 then receive 5x106 cells per infusion administered ID at study weeks 10, 14, 18, 22, 26, 30, 34, 38, 42, 46 and 50.
  Arms: Treatment Arm A
Biological: hTERT mRNA DC — Subjects receive 1x107 cells per infusion administered ID at study week 1, 2, 3, 4, 5, 6 then receive 1x107 cells per infusion administered ID at study weeks 10, 14, 18, 22, 26, 30, 34, 38, 42, 46 and 50.
  Arms: Treatment Arm B

SUMMARY:
The purpose of this research is to develop a new and powerful type of immune therapy for prostate cancer patients. This therapy involves vaccinations with special stimulator cells found in the human body called dendritic cells. These dendritic cells can take up proteins released from cancer cells and present pieces of these proteins to immune cells called T lymphocytes to create a strong stimulatory signal to fight the cancer.

One of these proteins is called telomerase, which is found on prostate cancers and is critically important for prostate cancer cells to grow. However, in most cancer patients, the immune system does not adequately destroy the tumor because the T cells are not stimulated sufficiently. T cells require strong stimulation before they grow and become active against cancer cells.

We have discovered that substances called ribonucleic acids (RNA), which carry the genetic instructions for the production of telomerase, can be used to overcome this problem and stimulate a strong immune response in cancer patients.

In order to test this hypothesis we have designed a clinical study and will enroll patients with metastatic prostate cancer expressing telomerase in order to determine whether or not this vaccine will stimulate T cells, which can recognize and kill prostate tumor cells.

The main objectives of this study are to find out whether injections with dendritic cells grown from blood cells and "pulsed" (mixed together for a short period of time) with RNA derived from the patient's own tumor are:

1. Safe without inducing any major side effects.
2. And effective in boosting the patient body's immunity against telomerase expressing prostate cancer cells.
3. Finally, we will test whether or not tumor shrinkage based on serum PSA levels or on X-ray studies will occur.

We hope that this new form of immune therapy, although in its infancy, will ultimately slow down tumor growth and prolong survival of prostate cancer patients.

DETAILED DESCRIPTION:
Primary objectives of trial include to evaluate the safety and biologic efficacy of hTERT mRNA transfected dendritic cells (DC), applied in a prime-boost format, to stimulate hTERT-specific CD4+ and CD8+ T-cell responses in subjects with metastatic prostate cancer. Secondary objectives include estimating objective clinical response, the duration of such responses, progression-free survival and overall survival among all subjects. The hTERT mRNA-transfected DC vaccine platform has previously been studied in several phase I/II trials and has demonstrated safety and bioactivity in subjects with metastatic prostate and renal cell carcinomas. The objective of this trial is to enhance the observed bioactivity of the vaccine by using a prime-boost strategy. This is an open label, uncontrolled safety and efficacy study. Subjects with metastatic prostate cancer will be eligible for this study and will receive 1x107 cells administered ID at study week 1,2,3,4,5, and 6 (Prime). Thereafter, subjects will be randomized with equal probability to receive either 5x106 cells administered ID at study week 10 followed by monthly immunizations (Treatment arm A) or 1x107 cells administered ID at study week 10 followed by monthly immunizations (Treatment arm B). The safety, biologic and clinical efficacy of each regimen will be analyzed. The study will be solely conducted at the University of Florida in Gainesville, FL. Subjects will be recruited through the oncology clinics of the Departments of Urology and Radiation Oncology. The vaccine will be manufactured in a dedicated GMP-compliant cell production facility located on the 4th floor of the Cancer Genetics Research Institute. Immunological testing will be performed in the Immunological Monitoring Core laboratory of the Department of Urology using standardized assay systems. Subjects with histologically or clinically confirmed metastatic prostate cancer (stages pT1-4, N0-3, M+) are eligible for this study. Subjects treated with medical hormone ablative therapy (LHRH analogues or estrogens) should continue to receive LHRH analogues only. In subjects receiving nonsteroidal medical hormonal treatment (i.e. flutamide or bicalutamide) and who are experiencing a rising PSA, a 4 week period of observation will be required following the discontinuation of the nonsteroidal antiandrogen prior to study entry. Subjects will be excluded from study if they have received chemotherapy or other forms of immunotherapy in the 4 weeks prior to study entry. They must not have a history of autoimmune disease, serious intercurrent chronic or acute illness, pulmonary disease, active hepatitis, serologic evidence for HIV, or be receiving corticosteroid or immunosuppressive therapy. All subjects must be older than 18 years. This is a randomized phase II clinical trial, in which up to 36 subjects will be randomized with equal probability to one of the two treatment arms. The objective of this trial is to decide which of the two treatment regimens should be selected for further testing. Hence, the primary objective of this trial is to select the arm with the highest biologic response and the first ranked arm will be selected for further study in a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have histologically or clinically confirmed adenocarcinoma of the prostate with either:

* metastatic prostate adenocarcinoma, Stage (T1-4, N+, M0) or (T1-4, N0-3, M+) OR
* two documented rising PSA levels while maintained on LHRH analogues.

  * Subjects who are receiving nonsteroidal antiandrogen therapy must discontinue therapy for 4 weeks prior to study entry.
  * Karnofsky Performance Status (KPS) greater than or equal to 80%
  * Age ≥ 18 years
  * Adequate hematologic function with:
* WBC ≥ 3000 mm3
* hemoglobin ≥ 9 mg/dl
* platelets ≥ 100,000/mm3

  • Adequate renal and hepatic function with:
* serum creatinine < 2.5 mg/dl
* bilirubin < 2.0 mg/dl

  • Adequate coagulation parameters with:
* Prothrombin Time < 1.5 x control
* Partial thromboplastin time < 1.5 x control • Ability to understand and provide signed inform consent that fulfills Institutional Review Board guidelines.

Exclusion Criteria:

* Subjects who have received radiation therapy within 4 weeks of pretreatment evaluation. (There must be at least 12 weeks if prior therapy included 89-Strontium between any prior therapy and study entry.)
* Subjects who have received chemotherapy or biologic regimens within 4 weeks of pretreatment evaluation.
* Subjects who have received immunotherapy within 4 weeks of pretreatment evaluation.
* Subjects who have not recovered from radiation, chemotherapy, or immunotherapy toxicities.
* Subjects with either previously irradiated or new CNS (central nervous system) metastases. (Pre-enrollment head CT is not required.)
* Subjects with a history of autoimmune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Subjects with serious intercurrent chronic or acute illness such as pulmonary (asthma or COPD) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the P.I. to constitute an unwarranted high risk for investigational drug treatment.
* Medical or psychological impediment to probable compliance with the protocol.
* Concurrent second malignancy other than non-melanoma skin cancer, or controlled superficial bladder cancer. In the event of prior malignancies treated surgically, the subject must be considered NED (no evidence of disease) for a minimum of 3 years prior to enrollment.
* Presence of an active acute or chronic infection, including symptomatic urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology).
* Subjects on steroid therapy (or other immunosuppressive agents such as azathioprine or cyclosporine A) are excluded on the basis of potential immune suppression. Subjects must have had 4 weeks of discontinuation of any steroid therapy prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this trial is to evaluate the safety of a boosting regimen using immunizations with two distinct doses of hTERT mRNA DC. | 50 Weeks
  All subjects will receive 1x107 cells administered ID at study weeks 1, 2, 3, 4, 5, and 6. Subjects will subsequently be randomized with equal probability to receive hTERT mRNA DC at study weeks 10, 14, 18, 22, 26, 30, 34, 38, 42, 46, and 50 at one of the following doses:
  * 5x106 cells per infusion administered ID (Treatment arm A).
  * 1x107 cells per infusion administered ID (Treatment arm B).

SECONDARY OUTCOMES:
PSA-specific T cells from pre- and post-therapy PBMC samples | 50 Weeks
  To analyze the induction of PSA-specific T cells from pre- and post-therapy PBMC samples among subjects enrolled in both treatment arms.
Calculate progression-free survival if subject responds to therapy. | 50 Weeks
  To monitor eventual clinical responses as evidenced on clinical response criteria and calculate progression-free survival if subject responds to therapy.
overall survival | 50 Weeks
  To determine overall survival for all subjects at one-year of follow-up.